CLINICAL TRIAL: NCT02122991
Title: Cardiovascular, Cerebrovascular, and Cognitive Function in SCI
Brief Title: Cardiovascular, Cerebrovascular, and Cognitive Function in Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jill M. Wecht, Ed.D., Research Health Scientist, James J. Peters Veterans Affairs Medical Center
Other Study IDs: WEC-13-024; 01492 (Other: MIRB)
Record Dates: First submitted 2013-07-01; First posted 2014-04-25 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; autonomic dysreflexia; baroreceptor integrity; sympathetic integrity; vagal integrity; autonomic integrity; arterial stiffness; cognitive function; traumatic brain injury; cerebral blood flow
MeSH Terms: conditions — Spinal Cord Injuries; Autonomic Dysreflexia; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Able-Bodied Controls: Subjects must be between the ages of 30 and 64 years old, be English-literate and able to provide informed consent. They must score at least 20/60 minimum acuity in their worst eye on the Snell Eye Exam, and score at least 22 on the Montreal Cognitive Assessment. Subjects MUST NOT HAVE: an acute illness or infection, history of stroke, recent illicit drug abuse (<6 months), unstable/uncontrolled seizures, neurodegenerative disease, Severe Traumatic Brain Injury (as determined by TBI screening tool), any significant history of neurological disease/disorder, any significant systemic illness or unstable medical condition (uncontrolled diabetes, hypo- or hyperthyroidism, systemic cancer), history of schizophrenia or bipolar disorder or any active psychosis, or alcohol/substance abuse or dependence (<6 months).
- Spinal Cord Injury: Subjects must be between the age of 30 and 64 years old, be English-literate and able to provide informed consent. They must be at least 1 year from the date of their spinal cord injury. They must score at least 20/60 minimum acuity in their worst eye on the Snell Eye Exam, and score at least 22 on the Montreal Cognitive Assessment. Subjects MUST NOT HAVE: an acute illness or infection, history of stroke, recent illicit drug abuse (<6 months), unstable/uncontrolled seizures, neurodegenerative disease, Severe Traumatic Brain Injury (as determined by TBI screening tool), any significant history of neurological disease/disorder, any significant systemic illness or unstable medical condition (uncontrolled diabetes, hypo- or hyperthyroidism, systemic cancer), history of schizophrenia or bipolar disorder or any active psychosis, or alcohol/substance abuse or dependence (<6 months).

SUMMARY:
Increased life expectancy in individuals with spinal cord injury (SCI) present clinicians with the challenge of managing the secondary complications of SCI with the chronic diseases common in an aging population. Cardiovascular disease, cerebral vascular disease, and cognitive dysfunction are among the primary challenges facing clinicians in the treatment of an aging population. Cognitive dysfunction has been reported in upwards of 60% of the SCI population, which have been primarily attributed to concomitant traumatic brain injury or pre-morbid conditions. Identifying possible modifiable risk factors which contribute to the increased prevalence of cognitive dysfunction in the SCI population is of significant clinical relevance and cardiovascular and cerebrovascular disorders have emerged as possible contributors to the cognitive disorders in the general population. These risk factors include: physical inactivity, chronically low or high blood pressure (BP), reduced blood flow to the brain, arterial stiffening, and impaired nervous system regulation of the cardiovascular system. These risk factors are particularly prominent in the SCI population as they represent a model of profound inactivity, have trouble regulating blood pressure, and suffer impaired cardiovascular regulation from their injury. In addition, we've recently reported deficits in blood flow to the brain at rest and during cognitive tests; with results being further impaired in SCI with chronically low blood pressure. Therefore the goals of this project are to determine the influence of cardiovascular and cerebral vascular responses at rest and during cognitive testing on test performance in 80 individuals with SCI compared to 50 age-matched non-SCI controls. All potential subjects will undergo a rigorous two-part screening process which consists of an initial screening via telephone and a detailed, in-person screening. Eligible subjects will be invited to participate in a 3 hour laboratory visit during which their arterial stiffness, blood pressure, heart rate, respiration rate and, blood flow to the brain will be monitored at rest and during a comprehensive series of cognitive tests.

We hypothesize that blood pressure and cerebrovascular response to testing will account significantly for performance in cognitive testing that otherwise would have been attributable to SCI status.

DETAILED DESCRIPTION:
The cognitive test battery will consists of the tests listed below, administered in the order given. Each test will be scored according to the

1. California Verbal Learning Test (Total & SD?)
2. Controlled oral word association test
3. Symbol Digit Modalities Test (Oral version)
4. Trail Making Test (Oral version)
5. Stroop Test (W?, C?, CW?)
6. Digit Span (Forwards, Backwards, and Sequencing)
7. California Verbal Learning Test (LD? & Recognition?)
8. Letter-Number Sequencing
9. California Verbal Learning Test (LD Forced recognition?)
10. WASI-II Sub-tests (Vocabulary, Similarities, and Matrix Reasoning)

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 30 and 64 years old
* If SCI, the duration of injury must be greater than 1 year
* At least 20/60 minimum acuity in worst eye on the Snell Eye Exam
* A score ≥22 on the Montreal Cognitive Assessment
* English literate
* Able to provide informed consent

Exclusion Criteria:

* Acute illness or infection
* Documented history of:

  * Stroke
  * Recent illicit drug abuse (from medical chart, within the past 6-months)
  * Unstable or uncontrolled seizures
  * Neurodegenerative disease including Alzheimer's disease, Parkinson's disease, Huntington's disease
  * Severe TBI (identified by TBI screening tool)
* Any significant history of neurological disease/disorders:

  * Alzheimer's disease
  * Parkinson's disease
  * Vascular dementia
  * Huntington's disease
  * Pick's disease
  * Lewy Body Dementia
  * Frontotemporal dementia
  * Normal pressure hydrocephalus
  * Brain tumor
  * Progressive supranuclear palsy
  * Seizure disorder
  * Multiple sclerosis
* Any significant systemic illness or unstable medical condition, including:

  * Uncontrolled diabetes mellitus,
  * Uncorrected hypothyroidism or hyperthyroidism,
  * Systemic cancer.
* History of schizophrenia or bipolar disorder or any active psychosis
* Alcohol or substance abuse or dependence within the past 6 months (from medical record)

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 80 subjects with chronic SCI and 50 age-matched non-SCI controls will be recruited from out-patient clinics at the JJP VAMC and the Center of Excellence. This includes subjects who have completed various protocols in the Cardiovascular autonomic testing laboratory or patients referred by their physicians following routine physical examinations. Physicians will be informed of the inclusion and exclusion criteria for this study and will be able to provide us with the assurance that the patient is an appropriate candidate for the study and that he/she was willing to speak with the study coordinators.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure (mmHg) | Up to 2 years
  To determine change in systolic blood pressure from seated rest to seated cognitive testing in subjects with and without spinal cord injury.
Performance on tests of information processing (WAIS-IV and Digit Span) and working memory (SDMT) | up to 2 years
  To compere cognitive performance on tests of working memory and information processing in individuals with and without spinal cord injury.

SECONDARY OUTCOMES:
Cerebral Blood Flow Velocity (cm/second) from the middle cerebral arteries | Up to 2 years
  To determine change in cerebral blood flow velocity from seated rest to seated cognitive testing in subjects with and without spinal cord injury.

CONTACTS AND LOCATIONS:
Overall Officials: Jill M Wecht, Ed.D., Principal Investigator — JJPVAMC
Locations (1):
- James J Peters VA Medical Center, The Bronx, New York, United States